CLINICAL TRIAL: NCT00438880
Title: A Phase I/II Trial of CpG 7909, Rituximab Immunotherapy, and Y-90 Zevalin Radioimmunotherapy for Patients With Previously Treated CD20+ Non-Hodgkin Lymphoma
Brief Title: Agatolimod Sodium, Rituximab, and Yttrium Y 90 Ibritumomab Tiuxetan in Treating Patients With Recurrent or Refractory Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS0382; NCI-2009-01275 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LS0382 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2015-09

CONDITIONS: Adult Non-Hodgkin Lymphoma; Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Nodal Marginal Zone Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — ProMune; Indium; Rituximab; X-Rays; Photons; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): See Detailed Description
  Interventions: Drug: Agatolimod Sodium; Radiation: Indium In-111 Ibritumomab Tiuxetan; Other: Laboratory Biomarker Analysis; Procedure: Radionuclide Imaging; Biological: Rituximab; Procedure: Single Photon Emission Computed Tomography; Radiation: Yttrium Y-90 Ibritumomab Tiuxetan

INTERVENTIONS:
Drug: Agatolimod Sodium — Given IV
  Other Names: (3'-5')d(P-thio)(T-C-G-T-C-G-T-T-T-T-G-T-C-G-T-T-T-T-G-T-C-G-T-T) Tricosasodium Salt; CpG 7909; PF-3512676; ProMune
Radiation: Indium In-111 Ibritumomab Tiuxetan — Given IV
  Other Names: IDEC In2B8; IDEC-In2B8; In 111 Ibritumomab Tiuxetan; In 111 Zevalin; indium In 111 ibritumomab tiuxetan
Other: Laboratory Biomarker Analysis — Correlative study
Procedure: Radionuclide Imaging — Undergo imaging scans
  Other Names: nuclear medicine scan; radioimaging; Radionuclide Scanning; Scan; SCINTIGRAPHY
Biological: Rituximab — Given IV
  Other Names: BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar BI 695500; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; RTXM83
Procedure: Single Photon Emission Computed Tomography — Undergo imaging scans
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Radiation: Yttrium Y-90 Ibritumomab Tiuxetan — Given IV
  Other Names: IDEC-Y2B8; IDEC-Y2B8 monoclonal antibody; Y 90 Ibritumomab Tiuxetan; Y 90 Zevalin; Yttrium Y 90 Ibritumomab Tiuxetan; yttrium Y90 ibritumomab tiuxetan

SUMMARY:
RATIONALE: Biological therapies, such as agatolimod sodium, may stimulate the immune system in different ways and stop cancer cells from growing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Radiolabeled monoclonal antibodies, such as yttrium Y 90 ibritumomab tiuxetan, can find cancer cells and carry cancer-killing substances to them without harming normal cells. Giving agatolimod sodium together with rituximab and yttrium Y 90 ibritumomab tiuxetan may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of agatolimod sodium when given together with rituximab and yttrium Y 90 ibritumomab tiuxetan and to see how well it works in treating patients with recurrent or refractory non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of CpG 7909 that can be delivered in four doses (days 6, 13, 20, 27) for patients with relapsed CD20+ non-Hodgkin's lymphoma. (Phase I) II. To assess the toxicity of CpG 7909 when combined with rituximab and Y-90 Zevalin in patients with lymphoma. (Phase I) III. To assess the overall response rate (CR + PR) of this regimen in relapsed diffuse large B cell lymphoma. (Phase II) IV. To assess the toxicity of the treatment regimen in patients with relapsed diffuse large B cell lymphoma. (Phase II) V. To assess the time to progression and duration of response in patients with relapsed diffuse large B cell lymphoma. (Phase II)

SECONDARY OBJECTIVES:

I. To report the response rate (complete remission + complete remission unconfirmed + partial remission) in this patient population after CpG 7909, rituximab, and Y-90 Zevalin. (Phase I) II. To compare the biodistribution of In-111 Zevalin radioimmunoconjugate scans before and after CpG 7909. (Phase I) III. To determine the HAMA/HACA rate in patients treated with this regimen. (Phase I) IV. To determine if CpG 7909 when given in the context of rituximab and Y-90 Zevalin can stimulate immune effector cells in the blood and tumor tissue. (Phase I)

OUTLINE:

This is a dose escalation study of agatolimod sodium followed by a phase II study.

PHASE I (patients with relapsed, refractory, or residual CD20+ non-Hodgkin lymphoma [closed to accrual as of 10/29/07]): Patients receive rituximab IV on days 1, 8 and 15, agatolimod sodium IV over 2 hours on days 6, 13, 20, and 27, and yttrium Y 90 ibritumomab tiuxetan* IV over 10 minutes on day 15 in the absence of disease progression and unacceptable toxicity.

*NOTE: Patients receive indium In 111 ibritumomab tiuxetan IV over 10 minutes on days 1 and 8. Patients undergo whole-body gamma camera imaging, single-photon emission computed tomography/CT scans, and blood sampling after each dose of indium In 111 ibritumomab tiuxetan to determine biodistribution. If biodistribution is acceptable, patients receive yttrium Y 90 ibritumomab tiuxetan.

PHASE II (patients with relapsed, refractory, or residual diffuse large B-cell lymphoma): Patients receive agatolimod sodium at the MTD as determined in phase I. Patients receive rituximab and yttrium Y 90 ibritumomab tiuxetan as in phase I.

*NOTE: Patients receive indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 8. Patients undergo whole-body gamma camera imaging and blood sampling after each dose of indium In 111 ibritumomab tiuxetan to determine biodistribution.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* The following histologic types by REAL classification and International Working Formulation (IWF) when applicable (NOTE: Closed to accrual as of 10/29/07): Small lymphocytic lymphoma; Lymphoplasmacytoid lymphoma; Follicular center lymphoma, follicular grades 1, 2, and 3; Extranodal marginal zone B cell lymphoma of MALT type; Nodal marginal zone B cell lymphoma
* The following histologic types by REAL classification and International Working Formulation (IWF) when applicable: Diffuse large cell; Transformed lymphoma
* Less than 25% bone marrow involvement of cellular marrow with lymphoma as determined by bilateral bone marrow aspirate and biopsy (the percent involvement should be estimated by the hematopathologist using all of the biopsy material)
* There is no limit on the number of prior therapies (patients who have previously received rituximab are eligible)
* Bi-dimensionally measurable disease: The patients must have >= 1 lesion that has a single diameter of >= 2 cm
* Absolute neutrophil count >= 1500/mm^3
* Platelet count >= 150,000
* Total lymphocyte count < 5000/mm^3 only for patients with small lymphocytic lymphoma
* HGB >= 8
* Biopsy-proven relapsed, refractory, or residual CD20+ non-Hodgkin's lymphomas; previous biopsies =<6 months prior to treatment on this protocol will be acceptable as long as there has not been intervening therapy; if the patient has received therapy for NHL between the time of the last biopsy and this protocol, then a re-biopsy is necessary
* ECOG performance status (PS) 0, 1, or 2
* Expected survival >= 3 months
* Willingness to provide all biologic specimens as required by the protocol
* Total bilirubin =< 2 x ULN mg/dL (if abnormal, direct bilirubin =< 1.5 x ULN)

Exclusion Criteria:

* Prior myeloablative therapies with autologous or allogeneic bone marrow transplantation or peripheral blood stem cell support
* Prior radioimmunotherapy including Y-90 Zevalin or 131-Iodine anti-B1 antibody or Lym-1
* Presence of CNS lymphoma
* Serious non-malignant disease such as active infection or other condition which in the opinion of the investigator would compromise other protocol objectives
* Major surgery other than diagnostic surgery =< 4 weeks prior to registration
* Another active primary malignancy
* Known HAMA/HACA (Human anti-mouse or anti-chimeric antibodies)
* Myelodysplastic syndrome or marrow chromosomal changes suggesting myelodysplasia
* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, abstinence, etc.)
* Failed stem cell collection
* Marrow cellularity =< 15% (as determined on all bone marrow samples)
* Known to have lymphoma related to HIV or AIDS (these patients are excluded because it is unknown what effects prolonged B-cell depletion will have on these patient's immune system)
* G-CSF or GM-CSF therapy =< 1 week prior to study registration (pegylated filgrastim =< 3 weeks)
* Myelosuppressive chemotherapy =< 3 weeks prior to study registration (=< 6 weeks if rituximab, nitrosourea, or Mitomycin C)
* Skin rash (such as Stevens-Johnson's syndrome or toxic epidermal necrolysis) with prior rituximab therapy should not be entered on this study because of the risk of reoccurrence of that skin toxicity
* Abnormal renal function (serum creatinine > 2 mg/dL)
* Pre-existent clinical autoimmune or antibody mediated diseases, including systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, and autoimmune thrombocytopenia (patients that have no clinical symptoms of these diseases, but merely have previously detected antibodies are eligible)
* Received prior external beam radiation therapy to > 25% of active bone marrow
* Corticosteroid therapy at the time the patient enters the protocol; patients using prednisone or its equivalent for adrenal failure or using < 20mg of prednisone/day for other benign causes are accepted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-10; Primary Completion 2010-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Witzig, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I of this study opened 10/20/2004 and accrued 30 patients before closing 10/29/2007. Eight patients were accrued to the Phase II portion at the maximum tolerated dose established in Phase I.
Groups:
- Phase I: Phase I patients will receive the following treatment:
  * 250 mg/m^2 Rituximab IV on days 1, 8, and 15 of a 27 day cycle
  * 5 mCi (Indium-111), 1.6 mg Ibritumomab IV on day 1
  * 10 mCi (Indium-111), 1.6 mg Ibritumomab IV on day 8
  * CpG 7909 (Agatolimod Sodium) doses will be assigned in groups of 6 patients. Dose levels will escalate in each group until maximum tolerability is attained (starting at 0.08 mg/kg and sequentially escalating to 0.16 mg/kg, 0.32 mg/kg, 0.48 mg/kg). Doses will be taken day 6, 13, 20, and 27 of a 27 day cycle.
  * 0.4 mCi/kg Yttrium-90 Zevalin IV on day 15
- Phase II: Phase II patients will receive the following treatment:
  * 250 mg/m^2 Rituximab IV on days 1, 8, and 15 of a 27 day cycle
  * 5 mCi (Indium-111), 1.6 mg Ibritumomab IV on day 8
  * 0.48 mg/kg CpG 7909 (Agatolimod Sodium) doses will be taken day 6, 13, 20, and 27 of a 27 day cycle.
  * 0.4 mCi/kg Yttrium-90 Zevalin IV on day 15
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 30 | 8
Completed | 30 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants accrued to this study were analyzed for baseline characteristics
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 30 | 8 | 38
Age, Continuous [Median (Full Range); unit: years] | 60.5 [36 to 80] | 68.5 [42 to 83] | 62.5 [36 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 4 | 17
  Male | 17 | 4 | 21
Region of Enrollment [Number; unit: participants]
  United States | 30 | 8 | 38

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of CpG 7909 as Determined Using the Number of Participants With a DLT at Each Dose Level
Description: Participants will be treated in cohorts of 6 patients at each dose level of CpG 7909 (0.08 mg/kg, 0.16 mg/kg, 0.32 mg/kg, 0.48 mg/kg) and observed for at least 10 weeks post treatment. If at most one of the 6 patients experiences a dose limiting toxicity (DLT), a new cohort of 6 patients will be treated at the next higher dose level. A DLT for this study is defined as patients with one of the following:
  * Absolute neutrophil counts or platelet counts below 10*10^9/L for 14 days
  * Absolute neutrophil counts greater than 0.5 or less than 1*10^9/L
  * Platelet counts greater than 10 or less than 50*10^9/L for 28 days.
  * Any grade 3 non-hematologic toxicity not explainable by another obvious cause as assessed using the Common Terminology Criteria for Adverse Events (CTCAE) v3.0.
  We are reporting the number of DLTs at each of the dose levels. The maximum tolerated dose will be 0.48 mg/kg or the largest dose level where 1 or fewer participants reports a dose limiting toxicity.
Time Frame: at least 10 weeks post treatment up to 3 months.
Population: Only participants accrued to the Phase I portion of this study were used to determine the maximum tolerated dose.
Measure: Number; unit: participants
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 30 | 0
participants
  Dose Level 1: (.08 mg/kg), n=6 | 0 |
  Dose Level 2: (.16 mg/kg), n=6 | 1 |
  Dose Level 3: (.32 mg/kg), n=6 | 0 |
  Dose Level 4: (.48 mg/kg), n=12 | 1 |

2. Primary Outcome: Tumor Response
Description: Complete Response (CR):
  * No measurable or nonmeasurable disease.
  * No symptoms of Lymphoma.
  * Non-palpable spleen, if palpable at baseline.
  * Histologically negative bone marrow, if positive at baseline.
  * All nodes <1.5 cm in transverse diameter.
  Partial Response (PR):
  * greater than 50% decrease from baseline in the sum of the products of the longest perpendicular diameters of the six largest dominant lesions.
  * No new lesions
  We are reporting the number of participants that attained a status of CR or PR.
Time Frame: Evaluations occur every three months up to a year
Population: Participants accrued to the Phase I portion of this study were not used to analyze the Phase II primary endpoint.
Measure: Number; unit: participants
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 0 | 8
participants
  Complete Response (CR) |  | 1
  Partial Response (PR) |  | 0

3. Secondary Outcome: Progression-free Survival
Description: The Progression-free survival (PFS) is defined as the time from registration to progression or death due to any cause. The distribution of PFS will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 1 year from treatment start date
Population: Only participants accrued to the Phase II portion of the study were evaluated for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 0 | 8
months |  | 1.57 [1.22 to 3.42]

4. Secondary Outcome: Duration of Response
Description: Duration of response (DoR) will be calculated from the documentation of response until the date of progression in the subset of patients who respond.
Time Frame: Up to 1 year from treatment start date
Population: The duration of response was not analyzed due to a lack of more than one response.
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Phase I | Phase II
Serious Adverse Events (participants affected / at risk) | 14/30 | 5/8
Other Adverse Events (participants affected / at risk) | 30/30 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=30) | Phase II (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 7 (7) | 0 (0)
Neutrophil count decreased (Investigations) | 10 (11) | 1 (1)
Platelet count decreased (Investigations) | 12 (20) | 4 (7)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=30) | Phase II (N=8)
Hemoglobin decreased (Blood and lymphatic system disorders) | 19 (40) | 8 (15)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (5) | 1 (1)
Localized edema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 26 (63) | 4 (7)
Neutrophil count decreased (Investigations) | 23 (37) | 4 (5)
Platelet count decreased (Investigations) | 26 (34) | 5 (7)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes